CLINICAL TRIAL: NCT05182801
Title: Banana Flower Extract in the Efficacy Verification Program of Hair and Body Health Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TCI Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 21-041-A2
Record Dates: First submitted 2022-01-04; First posted 2022-01-10 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Hair Loss
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo sachet (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo sachet
- Banana flower extract sachet (Experimental)
  Interventions: Dietary Supplement: Banana flower extract sachet

INTERVENTIONS:
Dietary Supplement: Placebo sachet — Blank
  Arms: Placebo sachet
Dietary Supplement: Banana flower extract sachet — Happy Angel Banana Flower Extract sachet
  Arms: Banana flower extract sachet

SUMMARY:
To assess Banana flower extract supplement on hair and body health care

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged above 20 years old

Exclusion Criteria:

* Subject who is not willing to participate in this study.
* Patients with diseases of the skin, liver, kidney.
* Subjects who have known cosmetic, drug or food allergies, difficulty in digestive tract absorption or disorder.
* Female who is pregnant or nursing or planning to become pregnant during the course of the study.
* The students taught by the PI.
* Subjects who have wounds on the scalp and subjects who have used drugs to treat the scalp, received hair transplants or other scalp treatments within six months

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-08-17 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
The change of hair loss amount | Change from Baseline hair loss amount at 12 weeks
  Collected and measured the weight of loss hair
The change of hair density | Change from Baseline hair density at 12 weeks
  Take a picture and observe the hair density
The change of hair follicle strength | Change from Baseline hair follicle strength at 12 weeks
  Pull up the hair of the frontal bone, temporal bone and occipital bone (approximately 60 hairs/area) to assess the number of hair loss in each area

SECONDARY OUTCOMES:
The change of scalp gloss | Change from Baseline scalp gloss at 12 weeks
  Chroma Meter MM500 was utilized to measure scalp gloss
The change of scalp redness | Change from Baseline scalp redness at 12 weeks
  Chroma Meter MM500 was utilized to measure scalp redness
The change of scalp health | Change from Baseline scalp health at 12 weeks
  Soft Plus was utilized to measure hair diameter
The change of hair diameter | Change from Baseline hair diameter at 12 weeks
  Mitutoyo C/N293-100 was utilized to measure hair diameter
The change of dihydrotestosterone of blood | Change from Baseline hair diameter at 12 weeks
  Venous blood was sampled to measure dihydrotestosterone
The change of testosterone of blood | Change from Baseline testosterone at 12 weeks
  Venous blood was sampled to measure testosterone
The change of SRD5A1 gene expression of blood | Change from Baseline SRD5A1 gene expression at 12 weeks
  Venous blood was sampled to measure SRD5A1 gene expression
The change of AR gene expression of blood | Change from Baseline AR gene expression at 12 weeks
  Venous blood was sampled to measure AR gene expression
The change of TGF-β gene expression of blood | Change from Baseline TGF-β gene expression at 12 weeks
  Venous blood was sampled to measure TGF-β gene expression
The change of IGF-1 gene expression of blood | Change from Baseline IGF-1 gene expression at 12 weeks
  Venous blood was sampled to measure IGF-1 gene expression

CONTACTS AND LOCATIONS:
Locations (1):
- Chia Nan University of Pharmacy ＆ Science, Tainan, Taiwan